CLINICAL TRIAL: NCT02531451
Title: The Effects of COX-inhibiting Drugs on Skeletal Muscle Adaptations to Resistance Exercise
Brief Title: The Effects of COX-inhibiting Drugs on Skeletal Muscle Adaptations to Resistance Exercise in Healthy Adults
Acronym: NSAID2015
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tommy Lundberg, PhD, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2014-004872-47
Record Dates: First submitted 2015-08-19; First posted 2015-08-24 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Skeletal Muscle Mass Regulation
Keywords: Muscle mass; strength; NSAID; Ibuprofen; resistance exercise
MeSH Terms: interventions — Ibuprofen; Aspirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ibuprofen (Experimental): Resistance exercise 20 sessions during 8 weeks Daily consumption of 1200 mg ibuprofen (400 mg x 3) during 8 weeks
  Interventions: Drug: Ibuprofen
- Acetylsalicylic acid (Active Comparator): Resistance exercise 20 sessions during 8 weeks Daily consumption of 75 mg acetylsalicylic acid (75 mg x 1) during 8 weeks
  Interventions: Drug: Acetylsalicylic acid

INTERVENTIONS:
Drug: Ibuprofen
  Arms: Ibuprofen
Drug: Acetylsalicylic acid
  Arms: Acetylsalicylic acid

SUMMARY:
In this study, healthy human subjects (18-35 yrs) are be randomised to consume 1200 mg ibuprofen or 75 mg acetylsalicylic acid daily during a training period of 8 weeks. During these weeks, subjects perform 2-3 supervised strength training sessions (knee extensions). Before and after training, muscle volume is measured by MRI, and muscle strength is assessed by isokinetic and isoinertial ergometers. Muscle biopsies are obtained from m. vastus lateralis to study gene and protein expression of markers regulating muscle protein turnover and prostaglandin synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Considered healthy
* Moderately trained
* 18-35 yrs

Exclusion Criteria:

* Cardiovascular disease
* Impaired kidney or liver function
* Lower limb injury
* Pregnancy
* Ulcer or gastrointestinal upsets
* Previous reactions to use of NSAID

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in Quadriceps muscle volume | Baseline and after 8 weeks training
  Measured through MRI

SECONDARY OUTCOMES:
Change in muscle gene expression | Baseline, 4 weeks and after 8 weeks training
  Through quantitative PCR and microarray
Change in muscle protein expression | Baseline, 4 weeks and after 8 weeks training
  Through Western Blots
Change in Quadriceps muscle strength | Baseline and after 8 weeks training
  Measured in strength dynamometers

CONTACTS AND LOCATIONS:
Overall Officials: Tommy Lundberg, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Sweden